CLINICAL TRIAL: NCT04565626
Title: Impact of Additional Unsupervised Peddle Bike Physiotherapy on Acutely Hospitalized Medicine Inpatients: a Feasibility Study
Brief Title: Impact of Additional Unsupervised Peddle Bike Physiotherapy on Acutely Hospitalized Medicine Inpatients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 116450
Record Dates: First submitted 2020-09-02; First posted 2020-09-25 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Additional Weekend Physiotherapy
Keywords: weekend; physiotherapy; deconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive additional exercise by independent use of a peddle bike on the weekends. This is in addition to their usual physiotherapy
  Interventions: Other: Additional weekend physiotherapy
- Control (No Intervention): This arm will receive usual physiotherapy

INTERVENTIONS:
Other: Additional weekend physiotherapy — Patients randomized to intervention would receive a Medical Exercise Bike Pedal Exerciser Mini Peddler to allow for an additional 20 minutes a day of unsupervised physiotherapy both during the week and on weekends.
  Arms: Intervention

SUMMARY:
During an acute hospitalization, deconditioning from decreased mobility can lead to functional decline. Muscle weakness can lead to frailty, which is linked to falls, immobility, rehospitalisation, institutionalization, and mortality. Many elderly do not regain muscle mass similar to prior to hospitalization and are discharged with worse than baseline function. Early mobilization and physical rehabilitation can improve or prevent loss of function in hospitalized patients. Weekend physiotherapy ensures gains made in mobility during the week are maintained, however, the benefit of additional weekend physiotherapy on acutely hospitalized Internal Medicine adult patients remains unclear.

Given this uncertainty, the investigators propose a randomized controlled trial pilot study to examine the outcomes of additional unsupervised physiotherapy. Patients randomized to intervention would receive a Medical Exercise Bike Pedal Exerciser to allow for an additional 20 minutes a day of un-supervised physiotherapy both during the week and on weekends.

Deconditioning will be measured for all study participants while hospitalized. After hospital discharge, patients will be telephoned on post-discharge day 3, to assess patient satisfaction and quality of life, and post-discharge day 30 to collect data regarding clinical outcomes (ER visits, re-hospitalizations, and falls).

The investigators hypothesize that it is feasible and safe to have additional unsupervised physiotherapy in the elderly population hospitalized for an acute illness on a medical ward and that this will result in improvement in function at discharge due to decreased hospital acquired deconditioning with improved mobility, quality of life and subsequent decreased readmission for falls.

DETAILED DESCRIPTION:
After obtaining written informed consent from eligible patients, study staff will randomize patients, collect demographics and hospital admission details from patients' hospital charts, and complete the Charlson Comorbidity Index (CCI) for all patients. The CCI will be completed using information gathered from patients' hospital chart. They will then perform the Barthel Index (BI) and Short Physical Performance Battery (SPPB) to determine a baseline physical ability of the patient.

The BI measures the extent to which patients can function independently and has mobility in their activities of daily living (ADL). The SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests (Guralnik et al., 2000). It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The Charlson Comorbidity Index categorizes and scores the comorbidities of patients. The CCI can be used to predict short term and long-term outcomes such as function, hospital length of stay and mortality rates.

The target sample size will be 75. This will be divided between intervention and no intervention (control). Patients will be allocated to either intervention with peddle bike for additional unsupervised exercise or current standard of care as control group. Randomization will be done using RedCap.

Patients randomized to intervention would receive a Medical Exercise Bike Pedal Exerciser Mini Peddler to allow for an additional 20 minutes a day of un-supervised physiotherapy both during the week and on weekends. Patients would be provided with an information pamphlet on the benefits of staying active during a hospitalization. Each bike will have an LCD monitor to keep track of patient use. They will receive a short teaching session on how to properly use the bike and record their use in their log. Exercise time (in minutes), distance (in kilometers) and calories will be recorded off the bike LCD monitor after each session and recorded in the patient's daily exercise log. They will also be assisted with follow-up meetings with the research therapist, and the involvement of the family (if available) from the outset, which has previously been shown to improve compliance. Patients randomized to the Bike Pedal Exerciser intervention will be assessed daily by the study staff & the medical team to ensure patients remain safe for use of the bike.

All participants (both intervention and control) will receive a Stepwatch to monitor their activity. This will be worn at all times in the study with the purpose to measure overall activity between the two groups. The investigators will manually remove the activity of the peddle bike from their overall activity in the intervention group to give a baseline activity rate. This will be to monitor for baseline activity in both groups and ensure that the intervention participants are not substituting the peddle bike for usual daily activity.

Deconditioning will be measured for all study participants on study day 3 and study day 6 (or the day of discharge) using the Timed Up and Go (TUG) test and Short Physical Performance Battery. For the TUG, patients will be asked to stand up from a chair, walk three metres, turn around, and walk back to the chair and sit.

After hospital discharge the research staff will follow up with all patients for 2 brief telephone interviews. On day 3 after discharge, Patient Satisfaction surveys* will be conducted by to assess patient satisfaction with their experience with their hospital stay & Peddle Bike program. They will also conduct the European Quality of Life, 5 dimensions* (EQ-5D-5 L) instrument to assess quality of life. At 30 days after randomization, the research staff will contact patients to conduct a brief interview consisting of: a functional status assessment (Barthel Index) and to collect data regarding clinical outcomes (ER visits, re-hospitalizations, and falls). Each telephone interview is expected to last approximately 10 minutes.

Peddle bikes will remain in a patient's room for the duration of their hospitalization and/or enrollment and will be cleaned between patient use to decrease risk of contamination.

Patients are assessed daily by their medical team as part of their standard care when hospitalized. If the team flags the patient as being incapable of using the peddle bike safely (i.e. patient is delirious or aggressive), the patient will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Cognitively safe for participation
3. Anticipated to remain hospitalized ≥48 hours
4. Inpatient, admitted to Internal Medicine Unit at University Hospital
5. Able to understand and follow instruction in the English language
6. Patient is receiving physiotherapy treatment from an LHSC inpatient physiotherapist

Exclusion Criteria:

1. Contraindications to exercise safely (pre-existing illness or acute illness) identified by patient's medical team
2. Patient is non-ambulatory at baseline
3. Patient or SDM is not interested in participating in the study
4. Patient is incapable of providing consent and no SDM is available
5. Communication/ language barrier. Participants need to be able to communicate and follow verbal instructions in English. Information pamphlets and consent forms will be only in English language.
6. Palliation or terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to additional weekend physiotherapy by unsupervised peddle bike | 1 year
  The investigators will assess the feasibility of a larger randomized control trial during which acutely hospitalized Internal Medicine patients participate in unsupervised pedal bike exercise for additional physiotherapy in addition to usual weekday hour physiotherapy. The investigators will collect data on adherence to protocol through the use of patient log to track patient activity. This patient log will track minutes of use per week of the peddle bike.
Recruitment | 1 year
  Ease of recruitment through monitoring of recruitment rate, refusal rate, and retention rate.
Emergent Adverse Events | 1 year
  Adverse events will be monitored through measuring falls, new fractures, and reported musculoskeletal pain requiring treatment.
Patient Perceptions | 1 year
  Patient perception of the peddle bike protocol will measured through a questionnaire at post discharge follow-up.
Completeness | 1 year
  Completeness measured as number of missing outcome measures

SECONDARY OUTCOMES:
Deconditioning as measured by the Timed up and go score | 1 year
  This score will be measured on day 3 and 6 of admission. This score is measured in seconds with a minimum being 0 seconds and no upper limit. A lower score indicates a better outcome.
Discharge destination | 1 year
  Identify discharge destination (home, low level residential care, high level residential care, and acute hospital transfer)
Health related quality of life measured by the European Quality of Life, 5 dimensions (EQ-5D-5 L) instrument | 1 year
  The investigators will measure health-related quality of life at 3 days post discharge from hospital using the European Quality of Life, 5 dimensions score. A minimum score is 0 and a maximum is 100. A higher score indicates a better outcome.
Length of stay | 1 year
  Decrease length of stay of index hospitalization, measured via admission and discharge dates
Readmission | 30 days
  Measure rate of readmission 30 days post discharge for falls measured via follow up telephone call and emergency room documentation
Deconditioning as measured by the Discharge Barthal Index for Activities of Daily Living score | 1 year
  This score will be measured on admission and 30 days after discharge from hospital. The minimum score is 0 and the maximum is 100. A higher score indicates a better outcome.
Deconditioning as measured by the Short Physical Performance Battery score | 1 year
  This score will be measured on the day of admission, and on days 3 and 6 of admission. The minimum score is 0 and the maximum score is 12. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Western, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The IPD will only be shared within the research team consisting of Dr. Melanie Le May, Dr. Erin Spicer, Dr. Marko Mrkobrada, Stephanie Handsor, and Karen Broadhurst